CLINICAL TRIAL: NCT03703453
Title: The Use of Resuscitative Endovascular Balloon Occlusion of the Aorta (REBOA) as an Adjunct to Advanced Cardiac Life Support in Non-traumatic Cardiac Arrest: an Early Feasibility Trial
Brief Title: Resuscitative EndoVascular Aortic Occlusion for Maximal Perfusion
Acronym: REVAMP
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, James I. Daley, Principal Investigator, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000023899
Record Dates: First submitted 2018-10-09; First posted 2018-10-12 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Cardiac Arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Intervention Model Description: REBOA in medical cardiac arrest patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- REBOA (Experimental): Patients undergoing REBOA for medical cardiac arrest
  Interventions: Device: ER-REBOA catheter

INTERVENTIONS:
Device: ER-REBOA catheter — The ER-REBOA™ catheter is a device that has been gaining increased use in the setting of severe trauma for the purposes of stopping intra-abdominal hemorrhage. The catheter is advanced through a femoral artery sheath into the aorta, where a balloon at its tip is inflated, occluding all distal blood flow (and stopping any hemorrhage while the patient can be prepared for definitive operative intervention).

SUMMARY:
REBOA is an endovascular technique that is becoming more widely used in the setting of severe trauma. It is a procedure where one uses the seldigner technique to advance a balloon tipped catheter into the femoral artery and then into the aorta. The balloon is then inflated to fully occlude blood flow to the distal aorta.

Study investigators hypothesize that this technique may be of use in the setting of medical cardiac arrest. By occluding the aorta and preventing distal blood flow during CPR, physicians might maximize perfusion to the heart and the brain, and promote return of spontaneous circulation and neurologic recovery.

Investigators plan to conduct an IDE approved early feasibility study using the ER-REBOA catheter in five patients who are in cardiac arrest of medical (i.e. non-traumatic) etiology. The primary outcomes will be feasibility and safety. Secondary outcomes will focus on procedural performance, hemodynamic response to aortic occlusion, and patient-centered outcome variables. Investigators plan to expand the study to an additional 15 patients if, after the initial five patients, the risk-benefit profile remains favorable.

DETAILED DESCRIPTION:
The proposed study will assess the safety, feasibility, and efficacy of the use of the ER-REBOA™ catheter as a means of increasing cardio-cerebral perfusion in medical cardiac arrest patients. The ER-REBOA™ catheter is a device that has been gaining increased use in the setting of severe trauma for the purposes of stopping intra-abdominal hemorrhage. The catheter is advanced through a femoral artery sheath into the aorta, where a balloon at its tip is inflated, occluding all distal blood flow (and stopping any hemorrhage while the patient can be prepared for definitive operative intervention).

Dr. Daley (along with previous investigators) has hypothesized that by using the device to occlude distal blood flow during medical cardiac arrest, one might increase the perfusion to the brain and heart, maximizing the patient's chance for cardiac and neurologic recovery. Aortic occlusion for medical cardiac arrest is supported by robust pre-clinical literature, but has not yet been studied in humans.

The proposed study is divided into two phases, with a different primary outcome in each phase. Phase 1 of the study is expected to occur over a period of 1 year. Phase 2 expected duration is 1.5 years. Each phase of the study will require separate FDA/IRB approval. Enrollment will take place at Yale-New Haven Hospital in New Haven, CT, the primary site for Phase 1 and Phase 2 of the study. A potential secondary site, the University of California, Davis, has been approved for trial participation but will not contribute to enrollment during Phase 1.

Phase 1 will primarily examine the feasibility and safety of the use of the ER-REBOA catheter in five non-traumatic cardiac arrest patients. If deemed feasible and safe, the PI will request permission from the FDA and the IRB to expand the study to Phase 2. Phase 2 will consist of the enrollment of a subsequent 15 patients (20 in total for both phase 1 and 2) with a primary focus on procedural performance, hemodynamic response to aortic occlusion, and patient-centered outcome variables. Per our hypothesis, if the ER-REBOA catheter is efficacious in medical cardiac arrest patients, an increase in systolic and diastolic blood pressure should be evident after the inflation of the intra-aortic balloon. Phase 2 will utilize the built in continuous arterial blood pressure monitoring capabilities of the device to assess for a significant blood pressure increase after the deployment of the aortic balloon.

ELIGIBILITY:
Inclusion Criteria

* The patient must have had a witnessed cardiac arrest2 of suspected medical etiology
* CPR initiation within approximately 6 minutes of collapse (as estimated based on history provided by EMS), either by EMS, hospital personnel, or a bystander

Exclusion Criteria

* Known active terminal illness or severe dementia
* Known aortic disease
* Age 80 or older
* Total resuscitation time greater than approximately 45 minutes (from start of CPR)
* Age less than 18
* Wards of the state
* Known or suspected (by physical exam or history) pregnancy
* Suspected traumatic cause of cardiac arrest
* Known Do Not Resuscitate (DNR) orders
* Anticipated difficult procedure (e.g. signs of peripheral vascular disease, severe obesity, or otherwise deemed likely to be difficult by enrollment staff)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-04-29 (Actual)

PRIMARY OUTCOMES:
Feasibility of aortic occlusion | The time expected for the procedure typically take between 10 and 15 minutes.
  The successful inflation of the aortic balloon at the level of the diaphragm with resultant occlusion of aortic blood flow. The procedure will be considered feasible if aortic balloons are deployed at the level of the diaphragm in at least 70% of patients attempted. The location of the balloon will be confirmed with bedside ultrasound and/or X-ray. Successful aortic occlusion will be confirmed using flow measurements on bedside ultrasound as well as detecting a lack of blood pressure distal to the aortic balloon using a pressure transducer in the femoral artery.
Safety of Procedure | Time of procedure to 90-days post-discharge
  Safety is defined by a composite prevalence of five pre-specified adverse events.
  •Composite events: blood vessel damage requiring intervention, arterial thromboembolism, lower extremity amputation, renal failure requiring non-temporary dialysis, lower extremity paralysis

SECONDARY OUTCOMES:
Time from first needle stick to sheath insertion | Time of micropuncture needle first insertion into common femoral artery until successful 7 French (Fr) sheath insertion into common femoral artery
  Procedural
Time from first needle stick to Resuscitative Endovascular Balloon Occlusion of the Aorta (REBOA) balloon inflation | Time when micropuncture needle first insertion into common femoral artery until REBOA catheter balloon successfully inflated with 8 cc saline
  Procedural
Number of needle sticks required for sheath insertion | Time from first micropuncture needle stick until successful insertion of 7 Fr sheath into common femoral artery up to 30 minutes
  Procedural
Change in systolic blood pressure after aortic occlusion | 1 minutes before and 15 minutes after aortic occlusion
  Hemodynamic
Change in diastolic blood pressure after aortic occlusion | 1 minute before and 15 minutes after aortic occlusion
  Hemodynamic
Change in end tidal carbon dioxide after aortic occlusion | 1 minute before and 15 minutes after aortic occlusion
  Hemodynamics
Change in oxygen saturation from pulse oximeter | 1 minute before and 15 minutes after aortic occlusion
  Hemodynamics
Change in coronary perfusion pressure | 1 minute before and 15 minutes after aortic occlusion
  Hemodynamics
Change in Electrocardiogram (ECG) patterns | 1 minute before and 15 minutes after aortic occlusion
  Hemodynamics
Neurologic function at 30 and 90 days | 30 and 90 days post enrollment
  Measured by Modified Rankin Scale (mRS) and Cerebral Performance Category (CPC).
  The mRS can help users determine the degree of disability in patients who have suffered a stroke or other causes of neurological disability by measuring the degree of disability or dependence in the daily activities of people. An mRS of a patient is compared over time to check for recovery and degree of continued disability. A score of 0 is no disability, 5 is disability requiring constant care for all needs; 6 is death. The mRS has been used in clinical research for over 30 years and is a common standard for assessing functional outcomes in patients. Multiple studies have shown that the mRS correlates with physiological indicators for neurological impairment.
  The CPC score is the most commonly used tool to assess this for both research and audit purposes. Most studies define a good outcome as a CPC score of 1 or 2, and a poor outcome (severe neurological disability, persistent vegetative state or
Rate of return of spontaneous circulation (ROSC) | Arrival in ED to sustained ROSC or death, assessed up to 1 hour
  Patient Oriented
Rate of Intensive Care Unit (ICU) Admission | Death in ED or admission to ICU post sustained ROSC, assessed up to 24 hours
  Patient Oriented
Length of stay in ICU and total length of hospitalization | Time of admission in ICU to discharge or death, assessed up to 90 days
  Patient Oriented

CONTACTS AND LOCATIONS:
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daley J, Morrison JJ, Sather J, Hile L. The role of resuscitative endovascular balloon occlusion of the aorta (REBOA) as an adjunct to ACLS in non-traumatic cardiac arrest. Am J Emerg Med. 2017 May;35(5):731-736. doi: 10.1016/j.ajem.2017.01.010. Epub 2017 Jan 12. PMID 28117180